CLINICAL TRIAL: NCT05259930
Title: Impact of Dietary Assessment and Intervention on Outcomes in Liver Cirrhosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Nualtra (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21143A01; 21/93 (Other: Beaumont Hospital Ethical Committee)
Record Dates: First submitted 2022-01-24; First posted 2022-03-02 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Sarcopenia; Cirrhosis, Liver
Keywords: branched-chain amino acid
MeSH Terms: conditions — Sarcopenia; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: Single Center randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chronic gastrointestinal disease (IBD and liver cirrhotic patients) (No Intervention): Liver cirrhotic patients to receive best practice nutritional assessment and supports
- branched-chain amino acid (BCAA) (Experimental): Liver cirrhotic patients to receive best practice nutritional assessment and supports in addition to a 12-week course of BCAA supplementation
  Interventions: Other: Amino MP9
- Healthy Control (No Intervention): Controls attending gastroenterology outpatient or endoscopy services with no chronic inflammatory GI disease.

INTERVENTIONS:
Other: Amino MP9 — Name used by Nualtra for their product of BCAA
  Arms: branched-chain amino acid (BCAA)

SUMMARY:
Malnutrition and reduced muscle mass have been associated with poor outcomes in many disease conditions including severe inflammatory bowel disease, liver failure and cancers. Studies have shown that use of an amino acid supplement can specifically support muscle and nutritional health of patients with liver cirrhosis and malnutrition in general. The investigators will perform new novel non-invasive measurements of muscle mass and strength as well as inflammatory markers and record food diaries in the investigators patients with inflammatory bowel disease, cirrhosis of the liver and other gastroenterology disease impacting patient nutrition. The investigators hope to determine if of the addition of BCAA in addition to best practice nutrition supports for patients with cirrhosis will improve muscle mass and clinical outcomes in the investigators patient cohort including hospitalization, rate of decompensations, frailty score and quality of life for patients with liver cirrhosis.

The investigators intend to investigate whether immune-metabolic profiles, circulating T-cells and circulating plasma cytokines (Afzal et al, J. Clin. Med. 2020) may act as biomarkers in combination with non-invasive novel markers of muscle mass in patients with chronic gastrointestinal illness, particularly cirrhosis to predict outcomes, and whether implementation of best practice nutritional supports with addition of Amino MP9 supplementation may impact functional outcomes. The immunometabolic profiles of these cohorts in relation to macrophage and T Cell function and differentiation have not been described previously.

The investigators also hope to develop a system facilitating accurate assessments of nutritional status in gastroenterology patients and determine if there is correlation with objective clinical activity measured using endoscopy, faecal calprotectin or radiological evidence of inflammation, currently measured as part of standard practice. Sub-analysis will investigate potential association between longitudinal diet evaluation using EDIP (empirical dietary inflammatory pattern) score and disease activity, clinical remission and response to medical therapy, all influencing quality of life and patient related outcome measures.

A prospective observational analysis of nutritional status and muscle mass or sarcopenia in patients attending gastroenterology services at Beaumont Hospital. Patients will be recruited from Gastroenterology and Hepatology outpatient clinics or inpatient capacity. Controls will be recruited from outpatient setting.

DETAILED DESCRIPTION:
The investigators objectives are summarised as,

Objective 1:

The investigators review 25-30 new patients, and approximately 120 return patients across 4 weekly clinics. These include approximately 40 patients with chronic liver disease or cirrhosis. In order to test validity of non-invasive markers of muscle mass including BIA device and thigh ultrasound in specific patient populations, the investigators propose recruitment of 100 patients and 30 controls.

Objective 2:

The investigators propose recruitment of 50 patients with cirrhosis to receive nutrition support plus Amino MP9 (BCAA supplementation), 50 patients with cirrhosis to receive nutrition support alone and 30 controls.

The following criteria are set for recruitment of patients into this study:

Inclusion Criteria

Confirmed cirrhosis (clinical or radiological diagnosis using liver biopsy, ultrasound/CT and/or transient elastography, Fibroscan) Age > 18 years Child Pugh score ≥B7 Active or recent (within the preceding 2 years) cirrhosis-related complication(s): including alcoholic hepatitis, ascites, variceal bleeding, spontaneous bacterial peritonitis, sepsis, encephalopathy, liver-related renal dysfunction, or hepatocellular carcinoma BCLC (Barcelona-Clinic Liver Cancer) stage A or B.

Exclusion Criteria

Active cancer (non-HCC) Advanced stage hepatocellular carcinoma (BCLC stage C or D) Pregnancy Breastfeeding/Lactation Lack of capacity for informed consent Hepatic Encephalopathy > Grade 2 at recruitment Listed for liver transplant Consumption of anabolic steroids for purpose of muscle development

In this study patients will divided recruited patients into 3 different arms, as follows:

Arm 1 (n=50): Patients with chronic liver disease and >F4 fibrosis on imaging (n=50) to receive best practice nutritional assessment and supports.

Arm 2 (n=50): Patients with chronic liver disease and >F4 fibrosis on imaging, to receive best practice nutritional assessment and supports in addition to a 12-week course of daily Amino MP9, BCAA supplement

Arm 3 (n=30): Controls attending gastroenterology outpatient or endoscopy services with no chronic inflammatory GI disease.

The investigators measurable outcomes includes:

Primary Outcome

1. Decompensation requiring hospital admission, surgery or medical intervention.
2. Improvement in anterior thigh muscle mass scores on ultrasound and non-invasive markers of muscle mass using SECA analysis

Secondary Outcome

1. Mortality
2. Impact of BCAA supplementation on immunometabolic markers in cirrhosis
3. Improvement in frailty and quality of life

Patients identified as suitable for recruitment will be invited to participate in this study which entails comprehensive nutritional assessment in addition to current standard medical practices and investigations {routine weight (in kg) and BMI(kg/m²)} at each hospital attendance. Patients with liver cirrhosis will be randomised 1:1 to receive either standard of care with nutrition assessment or nutrition assessment plus Amino MP9 supplementation. Patients in these groups and additionally, patients with chronic gastrointestinal diseases will undergo below assessments with regular dietetic analysis and review (currently not available due to resource limitations) to determine whether a prognostic score and cost benefit analysis of strict implementations of nutritional recommendations relates to prognosis. Completion at 0, 3, 12, 24 weeks.

Additional nutrition assessment offered will include:

1. Food frequency questionnaires (FFQ) (subsequent calculation of EDIP score)
2. Mid abdominal circumference measurement
3. Hand-grip strength
4. Sit-to-stand timed test
5. Mid-thigh circumference measurement
6. Gait speed test
7. Bilateral anterior thigh muscle mass via ultrasound
8. Muscle mass and strength through BIA device
9. Balance assessment

   * quality of life score assessment through CLD-Q questionnaire
   * For cirrhotic cohort the investigators will monitor level of encephalopathy through trail and stroop tests.

Immunometabolic Profile at at 0, 3, 12 and 24 weeks

-> Plasma cytokine (IL 1, 6, 8, 10, 23, 17, TNF), myostatin, leptin, ghrelin and adiponectin analysis. Immunometabolic circulating T-cell and macrophage profile

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cirrhosis (clinical or radiological diagnosis using liver biopsy, ultrasound/CT and/or transient elastography, Fibroscan)
* Age > 18 years
* Child Pugh score ≥B7
* Active or recent (within the preceding 2 years) cirrhosis-related complication(s): including alcoholic hepatitis, ascites, variceal bleeding, spontaneous bacterial peritonitis, sepsis, encephalopathy, liver-related renal dysfunction, or hepatocellular carcinoma BCLC (Barcelona-Clinic Liver Cancer) stage A or B.

Exclusion Criteria:

* Active cancer (non-HCC)
* Advanced stage hepatocellular carcinoma (BCLC stage C or D)
* Pregnancy
* Breastfeeding/Lactation
* Lack of capacity for informed consent
* Hepatic Encephalopathy > Grade 2 at recruitment
* Listed for liver transplant
* Consumption of anabolic steroids for purpose of muscle development

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Liver decompensation requiring hospital admission | 3 months
  Decompensated cirrhosis is defined as a patient with cirrhosis who presents with an acute deterioration in liver function that can manifest with the following symptoms:
  hepatic encephalopathy (equal or greater than 2), sepsis, new ascites/increase ascites, clinical jaundice, acute kidney injury according to modified RIFLE criteria and signs of gastrointestinal bleeding including melaena, haematemesis or coffee-ground vomiting
Liver decompensation requiring hospital admission | 6 months
  Decompensated cirrhosis is defined as a patient with cirrhosis who presents with an acute deterioration in liver function that can manifest with the following symptoms:
  hepatic encephalopathy (equal or greater than 2), sepsis, new ascites/increase ascites, clinical jaundice, acute kidney injury according to modified RIFLE criteria and signs of gastrointestinal bleeding including melaena, haematemesis or coffee-ground vomiting hepatic encephalopathy (equal or greater than 2), sepsis, new ascites/increase ascites, clinical jaundice , acute kidney injury according to modified RIFLE criteria and signs of gastrointestinal bleeding including melaena, haematemesis or coffee-ground vomiting
Anterior thigh muscle mass thickness | 3 months
  Improvement in anterior thigh muscle mass thickness on ultrasound (in millimetre)
Anterior thigh muscle mass thickness | 6 months
  Improvement in anterior thigh muscle mass thickness on ultrasound (in millimetre)
Segmental muscle mass | 3 months
  Improvement in segmental muscle mass analysis through Bio-impedance analysis device (SECA device). Muscle mass of arms, legs and trunk will be measured in kilogram.
Segmental muscle mass | 6 months
  Improvement in segmental muscle mass analysis through Bio-impedance analysis device (SECA device). Muscle mass of arms, legs and trunk will be measured in kilogram.

SECONDARY OUTCOMES:
Mortality | 6 months
Impact of BCAA supplementation on cytokines and immunometabolic markers in cirrhosis | 3 months
  Impact of BCAA on immune system this included measurements of (IL 1, 6, 8, 10, 23, 17, TNF), myostatin, leptin, ghrelin and adiponectin analysis. These will be measured with flow cytometry. Immunometabolic circulating T-cell and macrophage profile with flow cytometry. Measurements will be calculated with pg/mL scale.
Impact of BCAA supplementation on cytokines and immunometabolic markers in cirrhosis | 6 months
  Impact of BCAA on immune system this included measurements of (IL 1, 6, 8, 10, 23, 17, TNF), myostatin, leptin, ghrelin and adiponectin analysis. These will be measured with flow cytometry. Immunometabolic circulating T-cell and macrophage profile with flow cytometry. Measurements will be calculated with pg/mL scale.
Improvement in frailty | 3 months
  Improvement in frailty of liver cirrhotic patient and their quality of life based on liver frailty index { (-0.330 × gender - adjusted grip strength in kilogram) + (-2.529 × number of chair stands per seconds) + (-0.040 × balance time in second) + 6 }
Improvement in frailty | 6 months
  Improvement in frailty of liver cirrhotic patient and their quality of life based on liver frailty index { (-0.330 × gender - adjusted grip strength in kilogram) + (-2.529 × number of chair stands per seconds) + (-0.040 × balance time in second) + 6 }
Improvement in quality of life | 3 months
  Quality of life will be assessed with validated questionnaire, CLD-Q. This is consistent of 29 questions and it will assess patient's quality of life 2 weeks prior to assessments.
Improvement in quality of life | 6 months
  Quality of life will be assessed with validated questionnaire, CLD-Q. This is consistent of 29 questions and it will assess patient's quality of life 2 weeks prior to assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal College of Surgeons in Ireland, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
There is no consent or ethical approval for sharing IPD